CLINICAL TRIAL: NCT02607891
Title: A Phase 2, Double-blind, Randomized, Placebo-controlled Pharmacokinetic Trial in 2 Parallel Groups to Investigate Possible Drug-drug Interactions Between Stiripentol or Valproate and GWP42003-P in Patients With Epilepsy
Brief Title: A Study of Possible Drug-drug Interactions Between Stiripentol or Valproate and Cannabidiol in Patients With Epilepsy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GWEP1447 Blinded Phase; 2015-002939-18 (EudraCT Number)
Record Dates: First submitted 2015-11-16; First posted 2015-11-18 (Estimated); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Epilepsy
Keywords: Cannabidiol; GWP42003-P; Epidiolex; Stiripentol; Valproate
MeSH Terms: conditions — Epilepsy | interventions — Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- STP + GWP42003-P (Experimental): Administered orally, twice daily (morning and evening; immediately after the participant's STP dose), commencing with up-titration of 100 mg/mL GWP42003-P to a maintenance dose of 20 mg/kg/day over 11 days.
  Participants remain on the maintenance dose for a further 14 days. Dosing is tapered (10% each day) for participants who do not enter the open-label-extension (OLE) phase or who withdraw early.
  STP Arm: Last patient completion October 2018
  Interventions: Drug: GWP42003-P
- STP + Placebo (Placebo Comparator): Administered orally, twice daily (morning and evening; immediately after the participant's STP dose), commencing with up-titration of placebo to an equivalent maintenance dose of 20 mg/kg/day over 11 days.
  Participants remain on the maintenance dose for a further 14 days. Dosing is tapered (10% each day) for participants who do not enter the OLE phase or who withdraw early.
  STP Arm: Last patient completion February 2018
  Interventions: Drug: Placebo
- VPA + GWP42003-P (Experimental): Administered orally, twice daily (morning and evening; immediately after the participant's VPA dose), commencing with up-titration of 100 mg/mL GWP42003-P to a maintenance dose of 20 mg/kg/day over 11 days.
  Participants remain on the maintenance dose for a further 14 days. Dosing is tapered (10% each day) for participants who do not enter the OLE phase or who withdraw early.
  VPA Arm: Last patient completion February 2018
  Interventions: Drug: GWP42003-P
- VPA + Placebo (Placebo Comparator): Administered orally, twice daily (morning and evening; immediately after the participant's VPA dose), commencing with up-titration of placebo to an equivalent maintenance dose of 20 mg/kg/day over 11 days.
  Participants remain on the maintenance dose for a further 14 days. Dosing is tapered (10% each day) for participants who do not enter the OLE phase or who withdraw early.
  VPA Arm: Last patient completion January 2018
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GWP42003-P — Clear, colorless to yellow solution containing cannabidiol dissolved in the excipients sesame oil and anhydrous ethanol with added sweetener (sucralose) and strawberry flavoring.
  Other Names: Cannabidiol; CBD; Epidiolex
  Arms: STP + GWP42003-P; VPA + GWP42003-P
Drug: Placebo — Clear, colorless to yellow solution containing the excipients sesame oil and anhydrous ethanol with added sweetener (sucralose) and strawberry flavoring.
  Arms: STP + Placebo; VPA + Placebo

SUMMARY:
This trial consists of 2 parts: a double-blinded phase and an open-label extension phase. The blinded phase only will be described in this record. Participants will be randomized in a 4:1 ratio to receive GWP42003-P or matching placebo. The hypothesis is that levels of stiripentol (STP) or valproate (VPA) may be altered (increased or decreased) as a result of using GWP42003-P.

ELIGIBILITY:
Note: Participants who enroll in Sweden must be aged 18-55 years.

Key Inclusion Criteria:

* Participant must be taking STP (for the STP arm) or VPA (for the VPA arm) and no more than 2 other antiepileptic drugs (AEDs) during the blinded period of the trial.

  * In the VPA arm only, the participant must not be receiving STP (VPA allowed in STP arm).
* AED doses, including STP or VPA, must be stable for 4 weeks prior to screening and regimen must remain stable throughout the duration of the blinded period of the trial.
* Participant must have a documented magnetic resonance imaging/computerized tomography of the brain that ruled out a progressive neurologic condition.
* Participant must have experienced at least 1 countable uncontrolled seizure of any type (i.e., tonic-clonic, tonic, clonic, atonic, partial onset or focal: focal seizures with retained consciousness and a motor component, focal seizures with impaired consciousness, focal seizures evolving to bilateral secondary generalization) within 2 months prior to randomization.
* Intervention with vagus nerve stimulation and/or ketogenic diet must be stable for 4 weeks prior to baseline and the participant must be willing to maintain a stable regimen during the blinded period of the trial.
* Participant must abstain from alcohol during the blinded period of the trial.

Key Exclusion Criteria:

* Participant has clinically significant unstable medical conditions other than epilepsy.
* Participant has a history of symptoms related to a drop in blood pressure due to postural changes (e.g., dizziness, light-headedness, blurred vision, palpitations, weakness, syncope).
* Participant has a QT interval, corrected for heart rate with Bazett's formula (QTcB), greater than:

  * 450 msec for males.
  * 470 msec for females.
  * 480 msec if right bundle branch block is present.
* Participant has any history of suicidal behavior or any suicidal ideation of type 4 or 5 on the C-SSRS in the last month or at screening.
* Participant has had clinically relevant symptoms or a clinically significant illness in the 4 weeks prior to screening or enrollment, other than epilepsy.
* Participant is currently using felbamate and has been taking it for less than 12 months prior to screening.
* Participant has consumed alcohol during the 7 days prior to enrollment and is unwilling to abstain during the blinded phase of the trail.
* Participant is currently using or has in the past used recreational or medicinal cannabis, or synthetic cannabinoid-based medications (including Sativex®) within the 3 months prior to trial entry.
* Participant has any known or suspected history of any drug abuse or addiction.
* Participant is unwilling to abstain from recreational or medicinal cannabis, or synthetic cannabinoid based medications (including Sativex) for the duration for the study.
* Participant has consumed grapefruit or grapefruit juice 7 days prior to enrollment and is unwilling to abstain from drinking grapefruit juice within 7 days of pharmacokinetic visits.
* Participant has any known or suspected hypersensitivity to cannabinoids or any of the excipients of the Investigational Medicinal Product (IMP), e.g., sesame oil.
* Participant has received an IMP within the 12 weeks prior to the screening visit.
* Participant has significantly impaired hepatic function at the screening or randomization visit, defined as any of the following:

  * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 5 × upper limit of normal (ULN).
  * ALT or AST > 3 × ULN and total bilirubin (TBL) > 2 × ULN or international normalized ratio (INR) > 1.5.
  * ALT or AST > 3 × ULN with the presence of fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash, and/or eosinophilia (> 5%).

Ages: 16 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 35 (Actual)
Dates: Start 2016-11-09 (Actual); Primary Completion 2018-09-11 (Actual); Study Completion 2018-10-02 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) of STP, VPA, cannabidiol (CBD). | 0, 0.25, 0.5, 1, 1.5, 2, 4, 6, and 12 hours post-dose.
  The Cmax of STP, VPA and CBD is presented.
Time to the maximum plasma concentration (Tmax) of STP, VPA and CBD. | 0, 0.25, 0.5, 1, 1.5, 2, 4, 6, and 12 hours post-dose.
  The Tmax of STP, VPA and CBD is presented.
Area under the curve (AUC) from zero to final time of positive detection (0-t) of STP, VPA and CBD. | 0, 0.25, 0.5, 1, 1.5, 2, 4, 6, and 12 hours post-dose.
  The AUC(0-t) of STP, VPA and CBD is presented.
Area under the plasma concentration time curve over a dosing interval, where tau is the dosing interval [AUCtau]. | 0, 0.25, 0.5, 1, 1.5, 2, 4, 6, and 12 hours post-dose.
  The AUC(tau) of STP, VPA, and CBD is presented.

SECONDARY OUTCOMES:
Number of participants who experienced an adverse event. | Up to 11 weeks.
  The number of participants who experienced an adverse event during the trial is presented.
Number of participants with a clinically significant change in 12-lead electrocardiogram (ECG). | Up to 7 weeks.
  The number of participants with a clinically significant change in ECG is presented.
Number of participants with a clinically significant change in serum biochemistry. | Up to 7 weeks.
  The number of participants with a clinically significant change in serum biochemistry is presented.
Number of participants with a clinically significant change in hematology. | Up to 7 weeks.
  The number of participants with a clinically significant change in hematology is presented.
Number of participants with a clinically significant change in urinalysis. | Up to 7 weeks.
  The number of participants with a clinically significant change in urinalysis is presented.
Number of participants with a clinically significant change in vital signs. | Up to 7 weeks.
  The number of participants with a clinically significant change in vital signs (systolic blood pressure, diastolic blood pressure, pulse rate) is presented.
Number of participants with a clinically significant change in physical examination. | Up to 7 weeks.
  The number of participants with a clinically significant change in physical examination is presented.
Number of participants with a treatment-emergent suicidality flag. | Up to 7 weeks.
  Suicidality was assessed using the Columbia-Suicide Severity Rating Scale (C-SSRS). The number of participants with a treatment-emergent flag is presented.
Seizure frequency by subtype. | Up to 6 weeks.
  The frequency of each subtype of seizure at baseline and end of treatment is presented.
Number of participants with a treatment-emergent finding indicative of drug abuse liability. | Up to 7 weeks.
  Abuse liability was assessed through monitoring of triggering adverse events of interest and study medication accountability discrepancies. Any findings were assigned to an appropriate classification by the investigator. The number of participants with a treatment-emergent finding indicative of drug abuse liability is presented.
Cmax of 4-ene-VPA, clobazam (CLB), N-desmethylclobazam (N-CLB), levetiracetam (LEV), and topiramate (TOP). | 0, 0.25, 0.5, 1, 1.5, 2, 4, 6, and 12 hours post-dose.
  The Cmax of 4-ene-VPA, CLB, N-CLB, LEV, and TOP is presented.
Tmax of 4-ene-VPA, CLB, N-CLB, LEV, and TOP. | 0, 0.25, 0.5, 1, 1.5, 2, 4, 6, and 12 hours post-dose.
  The Tmax of 4-ene-VPA, CLB, N-CLB, LEV, and TOP is presented.
AUC(0-t) of 4-ene-VPA, CLB, N-CLB, LEV, and TOP. | 0, 0.25, 0.5, 1, 1.5, 2, 4, 6, and 12 hours post-dose.
  The AUC(0-t) of 4-ene-VPA, CLB, N-CLB, LEV, and TOP is presented.
AUC(tau) of 4-ene-VPA, CLB, N-CLB, LEV, and TOP. | 0, 0.25, 0.5, 1, 1.5, 2, 4, 6, and 12 hours post-dose.
  The AUC(tau) of 4-ene-VPA, CLB, N-CLB, LEV, and TOP is presented.

CONTACTS AND LOCATIONS:
Locations (5):
- SEIN - Epilepsy Institute in the Netherlands Foundation, Zwolle, Netherlands
- Spain (3):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Ruber Internacional, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ben-Menachem E, Gunning B, Arenas Cabrera CM, VanLandingham K, Crockett J, Critchley D, Wray L, Tayo B, Morrison G, Toledo M. A Phase II Randomized Trial to Explore the Potential for Pharmacokinetic Drug-Drug Interactions with Stiripentol or Valproate when Combined with Cannabidiol in Patients with Epilepsy. CNS Drugs. 2020 Jun;34(6):661-672. doi: 10.1007/s40263-020-00726-4. PMID 32350749